CLINICAL TRIAL: NCT01686594
Title: A Multi-center, Randomized Study on Oral 8-methoxypsoralen Plus UVA With or Without Maintenance Therapy in Mycosis Fungoides EORTC/ISCL Stage IA to IIB
Brief Title: PUVA Maintenance Therapy in Mycosis Fungoides
Acronym: M_PUVA_2012
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Peter Wolf, MD, Univ.Prof. Dr., Medical University of Graz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2012-000212-28; 24-169 ex 11/12 (Other: Ethics committee Medical University of Graz)
Record Dates: First submitted 2012-05-09; First posted 2012-09-18 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Patch/Plaque Stage Mycosis Fungoides
Keywords: Mycosis fungoides; Psoralen and UVA (PUVA); Photochemotherapy; Maintenance treatment; Immune function
MeSH Terms: conditions — Mycosis Fungoides | interventions — Methoxsalen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PUVA maintenance treatment (Active Comparator): Psoralen plus UVA (PUVA) treatment. The patients receive a standardized dose of oral 8-methoxypsoralen (Oxsoralen) 1 hour before UVA exposure
  Interventions: Drug: 8-methoxypsoralen
- No maintenance treatment (No Intervention): observation

INTERVENTIONS:
Drug: 8-methoxypsoralen — 8-methoxypsoralen 10mg per 20 kg body weight 1 hour before UVA exposure
  Other Names: Oxsoralen®; Gerot Pharmazeutika GmbH, Vienna, Austria
  Arms: PUVA maintenance treatment

SUMMARY:
The purpose of the study is to determine whether psoralen plus UVA (PUVA) photochemotherapy maintenance treatment prolongs disease-free survival of cutaneous T cell lymphoma (mycosis fungoides) patients.

DETAILED DESCRIPTION:
Background: Psoralen plus UVA (PUVA) photochemotherapy consists of the topical or oral application of psoralen, followed by exposure to UVA light. PUVA is used in various conditions, including early stages of mycosis fungoides (MF) and other primary and secondary lymphoproliferative disorders. PUVA has strong pro-apoptotic and immunomodulating properties, but the exact mechanisms by which PUVA leads to clearance of MF are not well understood. Although MF is generally a slowly progressing disease, it ultimately can spread to lymphoid tissues, peripheral blood, and other organs, leading to death.

Previous Work: PUVA therapy is a well-accepted first-line treatment option for skin-limited MF (stages IA, IB, and IIA), leading to complete remission in a high portion of patients (approximately 70 to 90%). Long-term remissions can be achieved with PUVA in a certain percentage of patients. However, in most cases MF lesions relapse after stop of PUVA after variable time intervals with a median time to relapse of 14 to 17 month, according to our own experience. Not only is little is known about the therapeutic mechanisms of PUVA in MF but as little is known about optimal duration and frequency of treatment (2, 3, or 4 times weekly), dose escalation, and maintenance therapy. Although PUVA has been introduced more than 30 years ago, there is lack of prospective controlled studies with clearly defined dose schemes and also an ongoing controversy whether PUVA maintenance therapy may prolong disease remission in MF upon initial complete clearance.

Hypothesis & Intended Work: We hypothesize that PUVA prolongs disease free survival in MF patients. In a randomized multicenter trial involving 9 centers in Austria, we plan to investigate (1) the clinical efficacy of PUVA and its maintenance therapy in MF and, (2) the mechanisms by which PUVA leads to disease clearance. In total, 82 patients will be enrolled and treated with a defined PUVA regimen with 2 exposures per week for 12 to 24 weeks. After 12 to 24 weeks of PUVA treatment, patients with complete remission will be randomized into two arms. In Arm A patients will be treated with PUVA maintenance therapy at constant single UVA doses. Maintenance treatment will be given once a week for one month (4 weeks), every 2 weeks for 2 months (8 weeks) and after three months once a month over 6 months. After 9 months of maintenance therapy patients will discontinue therapy. Patients in Arm B will receive no therapy. All patients will be followed until recurrence or at least 12 months (in non-recurrent patients) when the primary study analysis will be done. In addition, the follow-up will be extended to 60 months for long-term results.

The mechanistic action of PUVA will be studied by laboratory investigations, including immune function and cytokine analysis.

Outlook: A better understanding of the optimal regimen and the therapeutic mechanisms of PUVA in MF should help improving treatment strategies for this life-threatening disease. The understanding of the mode of action of PUVA in MF may also help to develop novel treatments using PUVA-affected pathways, allowing to achieve overall better long-term response and success.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically documented MF clinical stage IA-IIB (see Table1) confirmed by current or previous diagnostic lesion biopsy
* A Karnofsky performance score > 60
* No previous PUVA treatment
* Anti-ds-DNA (antinuclear antibodies) or anti-Ro/La antibodies: negative
* Acceptable organ function defined as follows:

SGOT (AST) and SGPT (ALT) < 2.5 times the upper limit of normal for the institution

* Creatinine < 2 times the upper limit of normal for the institution
* No evidence of severe cardiac insufficiency (NYHA grade III-IV)
* Women of child bearing potential must have a negative serum pregnancy test (ß-HCG) within seven (7) days prior to randomization
* Absence of any serious intercurrent illness or infection at time of entry into the study that could interfere with planned treatment
* Patients must be willing to accept limiting sun exposure on the day receiving PUVA treatment
* Written informed consent

Exclusion Criteria:

* Pregnancy and Lactation
* Photosensitive diseases such as lupus erythematosus or basal cell nevus syndrome
* Skin cancer syndromes such as xeroderma pigmentosum or basal cell nevus syndrome

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-02; Primary Completion 2018-07-02 (Actual); Study Completion 2018-07-02 (Actual)

PRIMARY OUTCOMES:
Recurrence after complete remission within 12 months post therapy | 12 months after end of therapy
  Recurrence is defined as mSWAT (modified severity weighted assessment tool ) >0.
  The primary outcome will be evaluated by survival analysis (log-rank test; Kaplan-Meier) comparing time to recurrence after complete remission between patients treated with maintenance therapy vs. patients without maintenance therapy.

SECONDARY OUTCOMES:
Quality of life | Week -4 to 0; week 12, 24, 36, and 48; month 15, 18, 21, 24, 36, 48, 60, and 72
  Compared to baseline
HADS | Week -4 to 0; week 12, 24, 36, and 48; month 15, 18, 21, 24, 36, 48, 60, and 72
  Hospital anxiety depression score, compared to baseline;
Cytokine response in serum | Week -4 to 0; week 6, 12, 24, and 48
  Compared to baseline
Levels of regulatory T cells | Week -4 to 0; week 6, 12, 24, and 48
  Compared to baseline
Function of regulatory T cells | Week -4 to 0; week 6, 12, 24, and 48
  Compared to baseline
Microscopic alterations | Week -4 to 0; and week 6; optional at week 12, 24, and 48; and in the follow-up from year 1 to 5
  Quantification of histologic response in skin biopsy
Cytokine expression in the skin | Week -4 to 0; and week 6; optional at week 12, 24, and 48; and in the follow-up from year 1 to 5
  Rt-PCR and immunohistochemical staining investigations

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wolf, MD, Principal Investigator — Medical University of Graz
Locations (9):
- Austria (9):
  - Medical University of Graz, Graz
  - Department of Dermatology, Medical University of Innsbruck, Innsbruck
  - Department of Dermatology, General Hospital of the City of Linz, Linz
  - Department of Dermatology, Hospital Salzburg - Paracelsus Private Medical University, Salzburg
  - Department of Dermatology, County Hospital St. Pölten, Sankt Pölten
  - Department of Dermatology, Medical University of Vienna, Vienna
  - Department of Dermatology, Hospital Hietzing, Vienna
  - Department of Dermatology, Klinikum Wels, Wels
  - Department of Dermatology, County Hospital Wiener Neustadt, Wiener Neustadt

REFERENCES:
- [Derived] Graier T, Fink-Puches R, Porkert S, Lang R, Pochlauer S, Ratzinger G, Tanew A, Selhofer S, Sator PG, Hofer A, Gruber-Wackernagel A, Legat FJ, Vieyra-Garcia PA, Quehenberger F, Wolf P. Quality of Life, Anxiety, and Depression in Patients With Early-Stage Mycosis Fungoides and the Effect of Oral Psoralen Plus UV-A (PUVA) Photochemotherapy on it. Front Med (Lausanne). 2020 Aug 5;7:330. doi: 10.3389/fmed.2020.00330. eCollection 2020. PMID 32850876
- [Derived] Vieyra-Garcia P, Fink-Puches R, Porkert S, Lang R, Pochlauer S, Ratzinger G, Tanew A, Selhofer S, Paul-Gunther S, Hofer A, Gruber-Wackernagel A, Legat F, Patra V, Quehenberger F, Cerroni L, Clark R, Wolf P. Evaluation of Low-Dose, Low-Frequency Oral Psoralen-UV-A Treatment With or Without Maintenance on Early-Stage Mycosis Fungoides: A Randomized Clinical Trial. JAMA Dermatol. 2019 May 1;155(5):538-547. doi: 10.1001/jamadermatol.2018.5905. PMID 30892603

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT01686594/Prot_SAP_000.pdf